CLINICAL TRIAL: NCT06406114
Title: Optimizing the Diagnostic Approach to Cephalosporin Allergy Testing
Acronym: DACAT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Kimberly Blumenthal, MD, MSc, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: 2024p000928; U01AI184071 (NIH)
Record Dates: First submitted 2024-04-17; First posted 2024-05-09 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Drug Allergy; Cephalosporin Allergy; Drug Hypersensitivity; Antibiotic Allergy; Beta Lactam Adverse Reaction; Drug-Induced Anaphylaxis; Cephalosporin Reaction
Keywords: Allergy; Antibiotic; Cephalosporin; Penicillin; Beta-lactam; Drug challenge; Skin testing; Adverse reaction; Anaphylaxis; Perioperative anaphylaxis
MeSH Terms: conditions — Drug Hypersensitivity; Hypersensitivity; Anaphylaxis | interventions — Monobactams; Cefazolin; Cefuroxime; Cefotaxime; Ceftazidime; Ceftriaxone; Cefepime; benzylpenicilloyl G polylysine; Penicillin G; Ampicillin; Histamine; Cephalexin; Cefaclor; Cefadroxil; Cefpodoxime; Cefdinir; Cefixime

STUDY DESIGN:
Intervention Model Description: The proposed study is a multi-site clinical trial of cephalosporin allergy diagnostic testing to determine the optimal diagnostic approach through unbiased assessments, including double-blind skin testing and double-blind placebo-controlled drug challenges using a crossover design.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Skin test reagents will be labeled blinded and prepared by a trained clinical trials pharmacy to maintain blinding. Drug challenges will be performed double-blind in a similar manner. The administrator, reader, and participant will all be blinded for each of these procedure types.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Similar cephalosporin first (Experimental): In visit 2, confirmed-allergic subjects will have a double-blind placebo-controlled drug challenge to a similar side chain cephalosporin, followed by a double-blind placebo-controlled challenge to a dissimilar side chain cephalosporin in visit 3. The randomization of which cephalosporin (similar or dissimilar side chain) is challenged in visits 2 and 3 differentiates the two arms.
  Interventions: Drug: Beta-lactam antibiotic (cefazolin, cefuroxime, cefotaxime, ceftazidime, ceftriaxone, cefepime, pre-pen, penicillin G, ampicillin, and histamine) double-blind skin testing; Drug: Culprit cephalosporin (cefazolin, ceftazidime, ceftriaxone, cefepime, cephalexin, cefaclor, cefadroxil, cefuroxime, cefpodoxime, cefdinir, or cefixime) double-blind placebo-controlled drug challenge; Drug: Similar cephalosporin (cefepime, ceftriaxone, cefaclor, cephalexin, cefixime, or cefdinir) antibiotic double-blind placebo-controlled drug challenge; Drug: Dissimilar cephalosporin (ceftriaxone or cefazolin) antibiotic double-blind placebo-controlled drug challenge; Drug: Amoxicillin double-blind placebo-controlled drug challenge
- Dissimilar cephalosporin first (Experimental): In visit 2, confirmed-allergic subjects will have a double-blind placebo-controlled drug challenge to a dissimilar side chain cephalosporin, followed by a double-blind placebo-controlled challenge to a similar side chain cephalosporin in visit 3. The randomization of which cephalosporin (similar or dissimilar side chain) is challenged in visits 2 and 3 differentiates the two arms.
  Interventions: Drug: Beta-lactam antibiotic (cefazolin, cefuroxime, cefotaxime, ceftazidime, ceftriaxone, cefepime, pre-pen, penicillin G, ampicillin, and histamine) double-blind skin testing; Drug: Culprit cephalosporin (cefazolin, ceftazidime, ceftriaxone, cefepime, cephalexin, cefaclor, cefadroxil, cefuroxime, cefpodoxime, cefdinir, or cefixime) double-blind placebo-controlled drug challenge; Drug: Similar cephalosporin (cefepime, ceftriaxone, cefaclor, cephalexin, cefixime, or cefdinir) antibiotic double-blind placebo-controlled drug challenge; Drug: Dissimilar cephalosporin (ceftriaxone or cefazolin) antibiotic double-blind placebo-controlled drug challenge; Drug: Amoxicillin double-blind placebo-controlled drug challenge

INTERVENTIONS:
Drug: Beta-lactam antibiotic (cefazolin, cefuroxime, cefotaxime, ceftazidime, ceftriaxone, cefepime, pre-pen, penicillin G, ampicillin, and histamine) double-blind skin testing — Percutaneous and intradermal skin testing will be performed in all participants. Concentrations for percutaneous testing; cefazolin (330 mg/ml), cefuroxime (90 mg/ml), ceftazidime (100 mg/ml), ceftriaxone (100 mg/ml), cefepime (200 mg/ml), pre-pen (undiluted), penicillin G (10,000 U/ml), ampicillin (20 mg/ml) and histamine (6 mg/ml). Concentrations for the first intradermal testing; cefazolin (3.3mg/ml), cefuroxime (1 mg/ml), ceftazidime (1 mg/ml), ceftriaxone (1 mg/ml), cefepime (2 mg/ml), Pre-PEN (undiluted), penicillin G (1000 U/ml), ampicillin (20 mg/ml), and histamine (0.1 mg/ml). Concentrations for the second intradermal testing; cefazolin (33mg/ml), cefuroxime (10 mg/ml), ceftazidime (10 mg/ml), ceftriaxone (10 mg/ml), cefepime (20 mg/ml), Pre-PEN (undiluted), penicillin G (10,000 U/ml), ampicillin (20 mg/ml) and histamine (0.1 mg/ml). Histamine and saline will be used as positive and negative controls.
Drug: Culprit cephalosporin (cefazolin, ceftazidime, ceftriaxone, cefepime, cephalexin, cefaclor, cefadroxil, cefuroxime, cefpodoxime, cefdinir, or cefixime) double-blind placebo-controlled drug challenge — After double-blind skin testing, participants will undergo a 3-step double-blind placebo-controlled drug challenge to their culprit cephalosporin (the cephalosporin they are suspected to be allergic to, either cefazolin, ceftazidime, ceftriaxone, cefepime, cephalexin, cefaclor, cefadroxil, cefuroxime, cefpodoxime, cefdinir, or cefixime). The challenges are 1:1 randomized to the order of active drug versus placebo. In Step 1, participants will receive 1:1000 of a full dose of either the culprit drug or placebo, followed by a 30-minute observation period. In Step 2, participants will receive 1:50 of a full dose of either, followed by another 30-minute observation period. In Step 3, participants are administered the full dose of either agent, followed by a 60-minute observation period. The same testing process is repeated for the second challenge.
Drug: Similar cephalosporin (cefepime, ceftriaxone, cefaclor, cephalexin, cefixime, or cefdinir) antibiotic double-blind placebo-controlled drug challenge — Participants will undergo a 3-step double-blind placebo-controlled drug challenge to a cephalosporin antibiotic that shares a similar side chain with their culprit. This will be cefepime for those allergic to ceftriaxone, cefaclor for those allergic to cephalexin, cefixime for those allergic to cefdinir, cefdinir for those allergic to cefixime, cephalexin for those allergic to cefaclor or cephadroxil, and ceftriaxone for those allergic to cefepime, cefuroxime, or cefpodoxime. The challenges are 1:1 randomized to the order of active drug versus placebo. In Step 1, participants will receive 1:1000 of a full dose of either the culprit drug or placebo, followed by a 30-minute observation period. In Step 2, participants will receive 1:50 of a full dose of either, followed by another 30-minute observation period. In Step 3, participants are administered the full dose of either agent, followed by a 60-minute observation period. The same testing process is repeated for the second challenge.
Drug: Dissimilar cephalosporin (ceftriaxone or cefazolin) antibiotic double-blind placebo-controlled drug challenge — Participants will undergo a 3-step double-blind placebo-controlled drug challenge to a cephalosporin antibiotic that has a dissimilar side chain to their culprit. This will be ceftriaxone for those allergic to cefazolin, and cefazolin for those allergic to any other cephalosporin. The challenges are 1:1 randomized to the order of active drug versus placebo. In Step 1, participants will receive 1:1000 of a full dose of either the culprit drug or placebo, followed by a 30-minute observation period. In Step 2, participants will receive 1:50 of a full dose of either, followed by another 30-minute observation period. In Step 3, participants are administered the full dose of either agent, followed by a 60-minute observation period. The same testing process is repeated for the second challenge.
Drug: Amoxicillin double-blind placebo-controlled drug challenge — Participants will optionally undergo a 3-step double-blind placebo-controlled drug challenge to Amoxicillin. The challenges are 1:1 randomized to the order of active drug versus placebo. In Step 1, participants will receive 1:1000 of a full dose of either the culprit drug or placebo, followed by a 30-minute observation period. In Step 2, participants will receive 1:50 of a full dose of either, followed by another 30-minute observation period. In Step 3, participants are administered the full dose of either agent, followed by a 60-minute observation period. The same testing process is repeated for the second challenge. The order of challenge to similar vs. dissimilar cephalosporin will be randomized as well.

SUMMARY:
Cephalosporin antibiotics are commonly used but can result in allergic reactions and anaphylaxis. There is no clear diagnostic approach for cephalosporin-allergic patients, and guidance for the use of other antibiotics in allergic patients is based on side chain chemical similarity and limited skin testing evidence. This project includes a clinical trial and mechanistic studies to optimize the approach to cephalosporin allergy and advance future diagnostics.

DETAILED DESCRIPTION:
Background:

In the United States, beta-lactam antibiotics are the leading cause of allergic reactions. Cephalosporin antibiotics, in particular, are the most common cause of drug-induced anaphylaxis and perioperative allergy. For penicillin allergy, the mechanism of allergy and the antigenic determinants are known; validated penicillin skin testing followed by drug challenge has a 100% negative predictive value to exclude an immunoglobulin (Ig)E-mediated reaction. For cephalosporin allergy, the antigenic determinants and mechanism are not known, and skin testing is not validated. The diagnostic test characteristics of skin testing with native cephalosporins remain unclear with no sensitivity nor specificity reported. Although beta-lactam cross-reactivity has been hypothesized to be from the similarity of the R1 side chains, rather than the beta-lactam ring, cross-reactivity estimates among beta-lactams vary. Furthermore, it is not known whether the variance in cross-reactivity is due to true allergy versus sensitization based on positive skin testing, given that drug challenges were not performed on skin-test-positive patients. While an IgE mechanism is assumed for cephalosporin allergy and supported by skin testing that has been positive, the biology has yet to be characterized, and some cephalosporin anaphylaxis can occur on the first exposure, which is inconsistent with an IgE mechanism. Given the complexity of cephalosporin structures and potential epitopes, there may be several distinct biologic pathways involved in cephalosporin allergy. Future diagnostics in cephalosporin allergy are reliant on determination of these biological pathways and finding key haptens.

Aims:

Current national practice guidelines related to cephalosporin allergy assessment are conditional and based on low-quality evidence. The overall goal is to identify the optimal diagnostic approach to cephalosporin allergy and determine beta-lactam cross-reactivity, while discovering the mechanism and antigenic determinants of cephalosporin allergy to advance future diagnostics. The investigators will do this through a clinical trial that will generate empirical evidence through novel trial procedures, double-blind skin testing, and double-blind placebo-controlled drug challenges. Specific aims are: 1) To determine the optimal approach to cephalosporin allergy evaluation; 2) To assess beta-lactam cross-reactivity in cephalosporin-allergic individuals; and 3) To investigate the antigenic determinants and mechanism of cephalosporin allergy.

Study Overview:

Enrolled and consented subjects will attend Visit 1 for baseline screening, sample collection, double-blind skin testing to a beta-lactam panel, and a double-blind placebo-controlled challenge to their culprit cephalosporin antibiotic. Results of the culprit cephalosporin challenge determine subject's study timeline. Subjects confirmed as non-allergic to their culprit cephalosporin will return for the End-of-Study Visit for venipuncture and blood collection, ending their participation in the study. Subjects who are confirmed as allergic to their culprit at Visit 1 will return for three additional visits; Visits 2 and 3 will include double-blind placebo-controlled challenges to a similar side chain and dissimilar side chain cephalosporin (as compared to the side chain of their culprit) to assess cross-reactivity. The order of these two challenges is randomized between Visit 2 and 3, and the order of whether a similar or dissimilar side chain cephalosporin is challenged first (in Visit 2) differentiates the comparator arms of this study. In Visit 4, subjects from both comparator arms will undergo a double-blind placebo-controlled challenge to a penicillin to assess cross-reactivity between cephalosporins and penicillins. After completion of this penicillin challenge, confirmed-allergic participants will return for an End-of-Study Visit. This visit will mark the end of their participation in the study. Venipuncture and sample collection will occur at each visit.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-70 years old.
2. Reaction history consistent with a potential immediate hypersensitivity reaction (pruritus, urticaria, erythema, angioedema, bronchospasm, wheezing, shortness of breath, anaphylaxis, or hypotension) to cefazolin, ceftazidime, ceftriaxone, cefepime, cephalexin, cefaclor, cefadroxil, cefuroxime, cefpodoxime, cefdinir, or cefixime.
3. English speaking or non-English speaking with translation services available.

Exclusion Criteria:

1. Severe concomitant medical condition (e.g., unstable coronary artery disease, congestive heart failure, severe chronic obstructive pulmonary disease, poorly controlled asthma, chronic renal failure, cirrhosis, or end-stage liver disease.)
2. History of Clostridioides difficile infection
3. Chronic spontaneous urticaria or systemic mastocytosis
4. Incident reaction required cardiopulmonary resuscitation
5. Reaction to 2 or more cephalosporin antibiotics
6. Active infection or antibiotic treatment within 7 days
7. Treatment with systemic antihistamines or corticosteroids within 7 days
8. Treatment with omalizumab or dupilumab within 60 days
9. Significant immunosuppression
10. Treatment with a beta-blocker or ACE inhibitor within 7 days
11. Use of investigational drugs within 60 days of participation
12. Anaphylaxis in the last 30 days
13. Penicillin anaphylaxis within the past year confirmed with positive penicillin skin tests
14. Prison or jail inmates, pregnant women, severe cognitive impairment
15. Current, diagnosed, mental illness or current, diagnosed, or self-reported drug or alcohol abuse that, in the opinion of the investigator, would interfere with the participant's ability to comply with study requirements
16. Past or current medical problems or findings from physical examination or laboratory testing that are not listed above, which, in the opinion of the investigator, may pose additional risks from participation in the study, may interfere with the participant's ability to comply with study requirements or that may impact the quality or interpretation of the data obtained from the study.
17. Inability or unwillingness of a participant to give written informed consent or comply with study protocol

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-05-05 (Actual); Primary Completion 2028-07-01 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with confirmed culprit cephalosporin allergy | Up to 7 weeks
  Placebo-controlled drug challenges will be used to confirm or disprove participant's cephalosporin allergies, and the proportion of included participants with confirmed allergies will be measured.
Cephalosporin skin test sensitivity and specificity | Up to 7 weeks
  Challenge results will be used as a reference standard to determine the sensitivity and specificity of cephalosporin skin testing.
Proportion of cross-reactivity to other cephalosporins in confirmed-allergic subjects | Up to 7 weeks
  The proportion of participants with confirmed cross-reactivity to dissimilar/similar cephalosporins than their culprit will be determined.

SECONDARY OUTCOMES:
Culprit cephalosporin skin test diagnostic characteristics | Up to 7 weeks
  The diagnostic testing characteristics of culprit cephalosporin skin tests will be evaluated, including positive predictive value (PPV), negative predictive value (NPV), and false positive rate.
Cephalosporin skin test diagnostic characteristic performance differences between risk groups | Up to 7 weeks
  Allergy history risk will be measured using a validated Drug Allergy History Tool. The PPV, NPV, and false positive rate of skin testing will then be compared through regression modeling to show differences in diagnostic characteristic performance between high-risk and low-risk groups.
Association between patient demographics and confirmed cephalosporin allergy | Up to 7 weeks
  Participant demographic traits will be collected and their associations with confirmed cephalosporin allergy will be presented as odds ratios with 95% confidence intervals.
Association between patient allergy history and confirmed cephalosporin allergy | Up to 7 weeks
  A validated Drug Allergy History Tool will be used to collect participant's allergy history, and associations of allergy history with confirmed cephalosporin allergy will be presented as odds ratios with 95% confidence intervals.
Proportion of nocebo responders | Up to 7 weeks
  The rate of nocebo response in those undergoing cephalosporin drug challenges will be measured.
Cephalosporin-specific antibody levels | Up to 54 months
  Cephalosporin drug- and hapten-specific antibody levels will be evaluated from serum using ELISA.
Cephalosporin-specific antibody binding | Up to 54 months
  Cephalosporin drug antibody binding epitopes will be presented using nanoallergens to evaluate rates of antibody binding and cell degranulation to gain a mechanistic understanding of cephalosporin allergy.

OTHER OUTCOMES:
Prevalence of nocebo response | Up to 7 weeks
  The prevalence of nocebo responses to drug challenges will be measured to understand how often these responses occur during cephalosporin challenges.
Graded severity of nocebo response reactions | Up to 7 weeks
  Respiratory, mucocutaneous, and cardiovascular symptoms and clinical presentation of nocebo response reactions will be collected and graded using the United States Drug Allergy Registry (USDAR) grading scale to determine the average severity of nocebo reactions. This scale is scored as either NR (no reaction) or values 0-4 indicating the severity of the reaction, with 0 being the mildest and 4 being the most severe.
Cephalosporin skin test clinical statistics | Up to 7 weeks
  The average diameter size of the wheal and flare during cephalosporin skin tests will be determined.
Tryptase levels in those with confirmed allergy | Up to 7 weeks
  In participants with confirmed cephalosporin allergy, tryptase levels will be evaluated and compared to determine if tryptase levels are associated with reaction grades.
Amoxicillin cross-reactivity in those with confirmed cephalosporin allergy | Up to 7 weeks
  Among those with confirmed cephalosporin allergy, the proportion with cross-reactivity to amoxicillin will be determined.
Amoxicillin skin test diagnostic characteristics in those with confirmed cephalosporin allergy | Up to 7 weeks
  Among those with confirmed cephalosporin allergy, the skin test diagnostic characteristics with amoxicillin will be determined, including positive predictive value (PPV), negative predictive value (NPV), and false positive rate.
Similar cephalosporin skin test diagnostic characteristics in participants with confirmed cephalosporin allergy | Up to 7 weeks
  Among those with confirmed cephalosporin allergy, the skin test diagnostic characteristics with a similar side-chain cephalosporin will be determined, including positive predictive value (PPV), negative predictive value (NPV), and false positive rate.
Dissimilar cephalosporin skin test diagnostic characteristics in participants with confirmed cephalosporin allergy | Up to 7 weeks
  Among those with confirmed cephalosporin allergy, the skin test diagnostic characteristics with a dissimilar side-chain cephalosporin will be determined, including positive predictive value (PPV), negative predictive value (NPV), and false positive rate.
Graded severity of cephalosporin allergic reactions | Up to 7 weeks
  Respiratory, mucocutaneous, and cardiovascular symptoms and clinical presentation of cephalosporin allergic reactions will be collected and graded using the United States Drug Allergy Registry (USDAR) grading scale to determine the average severity of cephalosporin reactions. This scale is scored as either NR (no reaction) or values 0-4 indicating the severity of the reaction, with 0 being the mildest and 4 being the most severe.
Proportion of delayed hypersensitivity reactions to cephalosporins | Up to 7 weeks
  The proportion of participants with delayed hypersensitivity reactions to cephalosporins will be recorded.
Incidence of adverse events with cephalosporin diagnostic tests | Up to 7 weeks
  The incidence rate of allergic and nonallergic adverse events (as graded by the United States Drug Allergy Registry (USDAR) grading scale [grades NR for no reaction and then grades 0-4 with four being the most severe reaction] and National Cancer Institute's Common Terminology Criteria for Adverse Events [grades 1 to 5, with grades 1 being the mildest and grade 5 being death]) in cephalosporin skin tests and drug challenges will be determined.

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly G Blumenthal, MD, MSc, Principal Investigator — Mayo Clinic; David A Khan, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (6):
- United States (6):
  - Mayo Clinic Arizona, Scottsdale, Arizona
  - University of California, San Francisco, San Francisco, California
  - Massachusetts General Hospital, Boston, Massachusetts
  - Rochester General Hospital, Rochester, New York
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Yes
Data will include demographics, clinical and procedure outcomes, and laboratory results. Investigators will preserve and share de-identified individual participant-level data (IPD) through submission to a controlled-access public repository. Investigators will apply the Safe Harbor method for de-identification of participant data. Participant informed consent forms will reflect this plan. To facilitate the use and interpretation of these data, the study protocol, data collection forms, case report forms, data dictionary, manual of operations, statistical analysis plan, and source code will be shared. Investigators will use Persistent Unique Identifiers (PIDs) to improve data findability across all dissemination outputs. PIDs used will include ORCID iDs for people, DOIs for outputs (e.g., datasets, protocols), and Research Resource IDentifiers (RRIDs) for resources. Investigators will also use indexed metadata to make scientific data easily findable.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: All scientific data generated from this project will be made available as soon as possible, and no later than the time of publication or the end of the funding period, whichever comes first. The duration of preservation and sharing of the data will be a minimum of 5 years after the funding period.
Access Criteria: Access to the data will be shared under controlled-access conditions as required by the policies of NIH/NIAID and the Mass General Brigham (MGB), which will serve as the sIRB. In accordance with HIPAA, scientific data derived from humans will be protected through de-identification, removal of information that may be used to infer the identity and shared under controlled-access conditions as required by NIH/NIAID and MGB institutional policy.